CLINICAL TRIAL: NCT07385391
Title: Development of a Novel Algorithm for Real-Time Bedside Assessment of Insulin Resistance in Critically Ill Patients Based on Continuous Glucose Monitoring Data: A Multicenter, Observational, Prospective Study
Brief Title: Development of a Novel Algorithm for Real-Time Bedside Assessment of Insulin Resistance in Critically Ill Patients Based on Continuous Glucose Monitoring Data
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: Insulin0114
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Metabolism Disorders; Insulin Resistance
Keywords: Metabolic Monitoring; Insulin Resistance; Prognosis
MeSH Terms: conditions — Critical Illness; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate a novel algorithm for the real-time assessment of insulin resistance in critically ill patients using Continuous Glucose Monitoring (CGM). Current methods for assessing insulin resistance are often invasive or unfeasible in the intensive care setting. By analyzing the dynamic correlation between CGM readings and reference blood glucose fluctuations, the investigators seek to construct a new algorithmic metric. The study will further evaluate the association of this new metric with established insulin resistance indices, organ function, and patient clinical outcomes.

DETAILED DESCRIPTION:
Insulin resistance (IR) is prevalent among critically ill patients, particularly those with sepsis, and is significantly associated with increased mortality, prolonged length of stay, and infectious complications. Consequently, real-time and accurate bedside monitoring of the degree of insulin resistance in this population is of paramount importance.

Current clinical modalities for assessing insulin resistance (IR) in critical illness remain insufficient. The "gold standard" hyperinsulinemic-euglycemic clamp (HEC) is restricted by invasiveness, complexity, and cost, while its artificial steady-state fails to reflect glucose dynamics under acute stress. Alternatively, HOMA-IR is a static, hepatic-focused measure; its reliance on fasting baselines is often unfeasible due to continuous nutrition, precluding accurate assessment of peripheral glucose disposal. Similarly, the Oral Glucose Tolerance Test (OGTT) is limited by gastrointestinal dysmotility and confounded by stress-induced insulin dysregulation. Consequently, a novel strategy for real-time, dynamic, and bedside IR assessment is urgently required to overcome these limitations.

This study aims to develop a novel algorithm for the real-time, bedside assessment of insulin resistance utilizing continuous glucose monitoring (CGM) data. A primary focus is the evaluation of the capability of CGM to capture dynamic glycemic fluctuations; specifically, the correlation between the magnitude of change in reference blood glucose between time points and the concurrent change in CGM readings will be analyzed. Based on the concordance of these dynamic variations, a new algorithmic metric is to be constructed. Subsequently, the association of this metric with established insulin resistance indices, organ function, and patient prognosis will be investigated to validate its clinical utility as a minimally invasive tool for monitoring metabolic status in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years and < 80 years
* ICU stay ≤48 hours
* Expected ICU stay > 24 hours
* APACHE II score≥ 8

Exclusion Criteria:

* local infection within the sensor placement area
* Laparotomy within lower abdomen
* Participated in this study before
* In other clinical trails

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patient
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | From date of study enrollment until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 60 days
  The incidence of all-cause death during the patient's stay in the Intensive Care Unit

SECONDARY OUTCOMES:
Incidence of Hyperglycemia | From date of study enrollment until ICU discharge, assessed up to 30 days.
  The proportion of participants who experience at least one episode of hyperglycemia during the observation period. Hyperglycemia is defined as a blood glucose level greater than 180 mg/dL (10 mmol/L).
Incidence of Hypoglycemia | From date of study enrollment until ICU discharge, assessed up to 30 days.
  The proportion of participants who experience at least one episode of hypoglycemia during the observation period. Hypoglycemia is defined as a blood glucose level less than 70 mg/dL (3.9 mmol/L). Severe hypoglycemia is defined as less than 40 mg/dL (2.2 mmol/L).
Duration of Vasopressor Dependency | From date of study enrollment until the date of vasopressor cessation for at least 24 hours, assessed up to 30 days.
  The total length of time a patient requires continuous intravenous vasoactive drugs to maintain adequate blood pressure.
Duration of Invasive Mechanical Ventilation | From date of study enrollment until the date of successful extubation, tracheostomy, or death from any cause, whichever came first, assessed up to 30 days
  The total length of time a patient requires endotracheal intubation and support from a mechanical ventilator.
Duration of Continuous Renal Replacement Therapy (CRRT) | From date of study enrollment until the date of CRRT discontinuation for at least 24 hours or death from any cause, whichever came first, assessed up to 30 days.
  The total length of time a patient requires continuous renal replacement therapy for acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, PhD, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China